CLINICAL TRIAL: NCT03056859
Title: Central Venous Catheterization in Obese Patients With Compass Device
Brief Title: Compass Device CVC Trial
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Collaborators: Centurion Medical Products (Industry)
Responsible Party: Principal Investigator, Neal Gerstein, Associate Professor, University of New Mexico
Other Study IDs: Compass Device Trial
Record Dates: First submitted 2017-02-14; First posted 2017-02-17 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Blood Pressure
Keywords: Operator satisfaction with device

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Enrolled Patients: Procedure: Central venous catheter placement with extravascular blood pressure transducer
  Interventions: Device: Extravascular blood pressure transducer

INTERVENTIONS:
Device: Extravascular blood pressure transducer — Listed device is included in central venous catheter placement apparatus for consenting patients, according to manufacturer directions
  Other Names: Compass Vascular Access

SUMMARY:
This is a single-arm observational trial of a device (Compass Vascular Access, Centurion Medical Products, Williamston MI). The device is a compact, sterile, single-use extravascular blood pressure transducer. This pressure measurement aids in confirmation of appropriate venous access. The investigators plan to enroll 40 consenting patients with BMI ≥35 who require central venous catheterization for clinical reasons independent of the existence of this study. The primary outcome is operator satisfaction.

DETAILED DESCRIPTION:
Forty (40) consenting patients meeting inclusion/exclusion criteria for this single-arm observational trial will be prepared as usual for central venous catheter (CVC) placement. The Compass pressure measurement device will be included in the CVC placement apparatus as per the manufacturer's directions. Data will be recorded on the placement procedure, operator satisfaction, routine patient demographics, and incidence of inadvertent arterial puncture.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥35

Exclusion Criteria:

* Pregnant women
* Adults unable to consent
* Non-English speakers
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at University of New Mexico main/adult operating rooms who require central venous catheter (CVC) placement for perioperative care.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Gerstein, MD, Principal Investigator — University of New Mexico School of Medicine
Locations (1):
- University of New Mexico Hospital, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified study data may be shared with other researchers, pending final decision by study PI and sponsor

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enrolled Patients
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [52 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 39.6 [36.2 to 43.2]

OUTCOME MEASURES:

1. Primary Outcome: Operator Satisfaction
Description: Operator satisfaction (0-10 scale; 0=totally dissatisfied, 10=totally satisfied)
Time Frame: 15 minutes
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 20
score on a scale | 8 [5 to 10]

2. Secondary Outcome: Arterial Puncture Incidence
Description: Incidence of arterial puncture
Time Frame: 15 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 20
Participants | 0

3. Secondary Outcome: Implement Used at Time of Arterial Puncture, if Any
Description: If arterial puncture occurred, list catheterization implement being manipulated at the time
Time Frame: 15 minutes
Population: There were no arterial punctures observed during the study.
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: One hour
Arm/Group | Enrolled Patients
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT03056859/Prot_000.pdf